CLINICAL TRIAL: NCT06237153
Title: Randomized Placebo Controlled Study of Triamcinolone Acetonide Extended Release Injection for Thumb (CMC) Osteoarthritis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Marie Badalamente (Other)
Responsible Party: Sponsor-Investigator, Marie Badalamente, Professor, Stony Brook University
Organization: Stony Brook University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Thumb 202; Thumb 202 (Other: stonyBrookU)
Record Dates: First submitted 2024-01-24; First posted 2024-02-01 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Carpometacarpal (CMC) Osteoarthritis
Keywords: Thumb Osteoarthritis
MeSH Terms: conditions — Capillary Malformations, Congenital, 1; Osteoarthritis

STUDY DESIGN:
Intervention Model Description: 30 patients randomly assigned to drug treatment or saline placebo injection (15 patients in each arm)
Who Masked: Participant, Investigator
Masking Description: Study coordinator holds randomization code.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Triamcinolone acetonide extended release suspension injection (Experimental): Active drug treatment
  Interventions: Drug: Triamcinolone Acetonide extended release suspension
- Saline Placebo Injection (Placebo Comparator): Placebo comparator
  Interventions: Drug: Triamcinolone Acetonide extended release suspension

INTERVENTIONS:
Drug: Triamcinolone Acetonide extended release suspension — Active steroid

SUMMARY:
The goal of this study is to investigate if a timed release steroid injection may be beneficial in treating carpometacarpal (CMC) joint (thumb) osteoarthritis. The main questions to be answered are:

1. does the steroid injection substantially reduce pain in the thumb
2. does the steroid injection help to increase thumb function Participants will be asked to undergo a thumb CMC joint injection and to attend follow up visits to assess pain and thumb function.

DETAILED DESCRIPTION:
Current Orthopaedic practice for CMC osteoarthritis involves prescribing thumb braces, oral non steroidal anti inflammatory medications (NSAID's) and/or corticosteroid injection(s) which may provide minimal relief, until symptoms become unbearable, leading to difficult and often complex surgical intervention and extended and painful post operative recovery times. Addition of a safe and effective and longer lasting conservative intervention may decrease pain and increase function in patients affected by CMC osteoarthritis.

Triamcinolone acetonide extended-release (TA-ER) suspension is novel and composed of polylactic-co-glycolic acid microspheres which allows for timed release of the steroid over the course of 12 weeks. It is FDA approved as Zilretta for injection and treatment of osteoarthritis of the knee.

We hypothesize that in a randomized, placebo controlled, double blind study that patients having TA-ER injection to the CMC joint will exhibit decreased pain levels and increased thumb function based on grip, tip and pinch strengths compared to placebo patients. One group of patients will receive CMC joint TA-ER injection and the other saline CMC joint injection. All will be followed for 12 weeks and one longer term follow up visit at 180 days.

Triamcinolone acetonide extended-release (steroid) injection for carpometacarpal (CMC) joint osteoarthritis may provide improved pain relief and thumb function as a conservative treatment for osteoarthritis of the base of the thumb.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female > 18 years of age.
2. X ray diagnosis of CMC osteoarthritis Eaton stages I, II or III.
3. VAS pain score in affected thumb of 5 or greater.
4. Written informed consent obtained from subject or subject's legal representative and ability for subject to comply with the requirements of the study.
5. Willing to abstain from use of the following protocol-restricted medications during the study to be kept in a log if non compliant.

   * Opioid or over the counter medications for pain for the study duration

Exclusion Criteria:

1. Females who are pregnant or nursing or plan to become pregnant during the study; women who plan to conceive during the study; or unwilling to practice birth control during participation in the study.
2. Presence of a condition or abnormality that in the opinion of the Investigator would compromise the safety of the patient or the quality of the data.
3. Known or suspected hypersensitivity to TA-ER (or component of TA-ER), triamcinolone acetonide.
4. Stage IV CMC osteoarthritis is excluded. Rationale for exclusion of stage IV is that these patients are most likely surgical candidates due to severe joint damage. Other exclusion criteria include rheumatoid arthritis, septic or gouty arthritis or psoriatic arthritis, thumb joint effusion, DeQuervain's disease, trigger thumb or history of CMC joint surgical reconstruction, or terminal or chronic and serious, uncontrolled associated medical conditions. Patients who have received hyaluronan or platelet rich plasma (PRP) injections to the affected CMC joint within 6 months will be excluded. Patients who have received a steroid injection to the affected CMC joint within 3 months will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-11-21 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Pain Score | Day 1 of injection to six months post injection
  PAIN

SECONDARY OUTCOMES:
QuickDash Thumb Function Questionnaire | Day 1 of injection to six months post injection
  Thumb Function
Grip Strength | Day 1 of injection to six months post injection
  Grip Strength
Pinch Strength | Day 1 of injection to six months post injection
  Pinch Strength
Key Strength | Day 1 of injection to six months post injection
  Key Strength

CONTACTS AND LOCATIONS:
Locations (1):
- Stony Brook Orthopaedics, Stony Brook, New York, United States

IPD SHARING:
Plan to Share IPD: No